CLINICAL TRIAL: NCT06426732
Title: The Trajectory of Blood Pressure During Pregnancy in Assisted Reproductive Females
Status: Recruiting | Type: Observational
Sponsor: The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Linlin Cui, Professor, The Second Hospital of Shandong University
Other Study IDs: 2022-919
Record Dates: First submitted 2024-05-18; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Natural pregnancy group
- Assisted Reproductive Technology Group

SUMMARY:
The incidence of gestational hypertension and preeclampsia in the assisted reproductive technology population during pregnancy was significantly higher than that in the general normal pregnancy population. The use of assisted reproductive technology in this population due to infertility is often accompanied by many hypertension-related factors. We established a prospective cohort study based on assisted reproductive technology pregnancy population and natural pregnancy population. Through continuous monitoring of blood pressure changes and other risk factors during pregnancy in the two groups, we explored the trajectory trend and inflection point of assisted reproductive technology pregnancy population blood pressure during pregnancy. Through factor analysis, the risk factors of elevated blood pressure during pregnancy can be clearly identified, so as to carry out early intervention and strengthen the control of risk factors of elevated blood pressure in assisted reproductive technology population, in order to expect benign maternal and infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

-Exposure group:

Mother: Seen in the obstetrics department of our hospital and meet the following conditions at the same time:

1. Complete at least one cycle of IVF or ICSI, PGD or IVM treatment (including natural cycles);
2. Clinical pregnancy was obtained after treatment. Offspring: Offspring born after in vitro fertilization-embryo transfer technique.

   * Non-exposed group:

Mother: A mother who conceived naturally. Offspring: 1) Offspring born by natural pregnancy. 2) Offspring born from natural pregnancy of exposed mothers.

Exclusion Criteria:

* Unwilling to participate in this research;
* Unable to participate in this study due to special reasons, such as death, immigration, loss to follow-up;
* Hereditary diseases, mental diseases, malignant tumors, pre-pregnancy hypertension, uterine malformations and other reproductive organ malformations;
* Pregnant women who voluntarily terminate pregnancy due to non-preeclampsia factors;

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: collect sixty patients in each group
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The Trajectory of Blood Pressure During Pregnancy in Assisted Reproductive Females | from pregnancy to delivery
  The Trajectory of Blood Pressure During Pregnancy in Assisted Reproductive Females

CONTACTS AND LOCATIONS:
Locations (1):
- Cui linlin, Jinan, China